CLINICAL TRIAL: NCT07030595
Title: A Randomized, Open-Label, Multi-Center, Phase 3 Study to Evaluate the Efficacy and Safety of AP301 on Serum Phosphorus Control in Chronic Kidney Disease Patients Receiving Maintenance Dialysis With Hyperphosphatemia
Brief Title: AP301 Efficacy and Safety in Chinese Dialysis Patients With Hyperphosphatemia
Acronym: RESPOND-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alebund Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP301-HP-02
Record Dates: First submitted 2025-06-05; First posted 2025-06-22 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-06

CONDITIONS: ESRD (End Stage Renal Disease); Chronic Kidney Disease(CKD); Hyperphosphatemia; Hyperphosphatemia in Chronic Kidney Disease; Dialysis; Chronic Kidney Disease, Receiving Dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia | interventions — Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AP301 (Experimental): A blood phosphate-lowering medication containing iron
  Interventions: Drug: AP301
- Sevelamer Carbonate (Active Comparator): A marketed blood phosphate-lowering medication
  Interventions: Drug: Sevelamer carbonate (Renvela®)
- AP301 Low Dose (Experimental): A blood phosphate-lowering medication containing iron, but with a low dose considered as ineffective
  Interventions: Drug: AP301 Low Dose

INTERVENTIONS:
Drug: AP301 — Three times a day, administered orally with three meals at a daily dose level from 2.1g to 9.1g
  Arms: AP301
Drug: Sevelamer carbonate (Renvela®) — Three times a day, administered orally with three meals at a daily dose level from 2.4g to 9.6g
  Arms: Sevelamer Carbonate
Drug: AP301 Low Dose — Three times a day, administered orally with three meals at a daily dose level of 0.375g.
  Arms: AP301 Low Dose

SUMMARY:
This Phase 3 clinical trial is the pivotal study of AP301 aiming to evaluate the efficacy and safety of AP301 for controlling serum phosphorus in chronic kidney disease receiving hemodialysis and peritoneal dialysis in Chinese patients with hyperphosphatemia.

DETAILED DESCRIPTION:
This study has two primary efficacy objectives. The primary efficacy objective 1 is to evaluate the superiority of maintenance dose versus low dose of AP301 on serum P control in dialysis patients with hyperphosphatemia. The primary efficacy objective 2 is to evaluate the non-inferiority of AP301 versus sevelamer carbonate on serum phosphorus control. Besides these two primary efficacy objectives, this study will also evaluate the serum phosphorus control equivalence and the safety for AP301 produced from two APIs (Active Pharmaceutical Ingredient) in the last 8 weeks of drug exposure.

Patients will start dosed after eligibility confirmation. The treatment period will last 52 weeks in total, including:

A) A 24-week sevelamer carbonate active control phase in which serum phosphorus level at the end of Week 12 will be measured for the analysis of primary efficacy endpoint 2, B) A 3-week AP301 low dose control phase in which serum phosphorus level at the end of Week 27 will be measured for the analysis of primary efficacy endpoint 1, and C) A 25 or 28-week extension treatment phase

The investigational treatments will be AP301. Sevelamer carbonate will be provided as active control in active control and extension treatment phase and AP301 125 mg as ineffective control in low dose control phase.

A) The starting dose of AP301 is one 700 mg capsule 3 times daily. The dosage is to be adjusted based on their serum phosphorus level and safety assessmentsevery two or four weeks. The maximal dose is to be 10 capsules daily.

B) The starting dose of sevelamer carbonate will be one to two 800 mg capsules 3 times daily. The dosage is to be adjusted based on their serum phosphorus level every and safety assessments two or four weeks. The maximal dose is to be 12 capsules daily.

Then, a 2-week safety observation will be followed after the last dosing.

ELIGIBILITY:
Key Inclusion Criteria:

* Provision of signed and dated ICF
* Adult when signing the ICF
* Patients on dialysis for ≥ 3 months before signing the ICF and throughout the study
* For HD patients, spKt/V ≥ 1.2; for PD patients, total Kt/V ≥ 1.7/week
* For patients who receive phosphate binders and their serum phosphate level is:

  1. Screening: 1.13 mmol/L (3.5 mg/dL) ≤ serum phosphate < 2.58 mmol/L (8.0 mg/dL)
  2. After washout: 1.94 mmol/L (6.0 mg/dL) ≤ serum phosphate < 3.23 mmol/L (10.0 mg/dL)
* For patients who do not receive phosphate binders over 2 weeks and their serum phosphate level is:

  1. Screening: 1.94 mmol/L (6.0 mg/dL) ≤ serum phosphate < 3.23 mmol/L (10.0 mg/dL)

Key Exclusion Criteria:

* History or plan of kidney transplantation
* History or plan of parathyroid intervention 6 months before signing the ICF
* Serum calcium < 1.9 mmol/L (7.6 mg/dL) or > 2.75 mmol/L (11 mg/dL) at screening
* Serum intact parathyroid hormone > 110 pmol/L (1000 pg/mL) at screening
* Presence of clinically significant gastrointestinal (GI) disorder
* History of gastrectomy or duodenectomy, or GI surgery within 3 months before signing the ICF
* Known allergic to any ingredient of AP301 or Sevelamer Carbonate, or known history of severe allergies leading to emergency medical care
* Female who are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Change in serum phosphorus levels between AP301 and AP301 low dose groups in hyperphosphatemic patients | From the end of Week 24 to the end of Week 27
  The serum phosphorus will be measured with a standard laboratory test. The change in serum phosphorus levels will be compared between the group receiving AP301 and the group receiving AP301 low dose.
Change in serum phosphorus levels between AP301 and sevelamer carbonate groups in hyperphosphatemic patients | From Baseline to the end of Week 12
  The serum phosphorus will be measured with a standard laboratory test. The change in serum phosphorus levels will be compared between the group receiving AP301 and the group receiving sevelamer carbonate.

SECONDARY OUTCOMES:
The achievement rate of serum phosphorus in the target range 1.13-1.78 mmol/L (3.5-5.5 mg/dL) (both inclusive). | From Baseline to the end of Week 52.
  The serum phosphorus will be measured with a standard laboratory test.
Changes in serum calcium | From Baseline to the end of Week 52
  The serum calcium in the blood will be measured with a standard laboratory test.
Changes in serum calcium times phosphorus product | From Baseline to the end of Week 52
  The serum calcium and phosphorus in the blood will be measured with standard laboratory tests.
Changes in intact parathyroid hormone | From Baseline to the end of Week 52
  The intact parathyroid hormone in the blood will be measured with a standard laboratory test.
Changes in serum bone-specific alkaline phosphatase | From Baseline to the end of Week 52
  The serum bone-specific alkaline phosphatase in the blood will be measured with standard laboratory tests.
Changes in osteocalcin | From Baseline to the end of Week 52
  The serum osteocalcin in the blood will be measured with a standard laboratory test.
Number of adverse events | From Baseline to Follow-up (up to 54 weeks)
Changes in serum iron parameters | From Baseline to the end of Week 52
  The serum iron parameters will be measured with standard laboratory tests.
Change in QT intervals measured by 12-lead electrocardiogram test over time | From Baseline to the end of Week 52
  The duration of QT intervals will be measured with a standard 12-lead electrocardiogram test.
Number of participants with abnormal vital signs | From Baseline to the end of Week 52
  The vital sign will consist of pulse rate and blood pressure with standard measurements.
Number of participants with abnormal laboratory tests results | From Baseline to the end of Week 52
  The laboratory tests will be measured with standard validated methods, involving hematology, biochemistry, bone markers, iron parameters and others.

OTHER OUTCOMES:
Changes in average serum phosphorus levels | From the end of Week 48 to the end of Week 52
  The serum phosphorus will be measured with a standard laboratory test.
Number of adverse events | From the end of Week 48 to the end of Week 52

CONTACTS AND LOCATIONS:
Locations (50):
- China (50):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Jilin Province People's Hospital, Jilin, Changchun
  - The Second Norman Bethune Hospital of Jilin University, Jilin, Changchun
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Dongguan People's Hospital, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - The First People's Hospital of Nanning, Nanning, Guangxi
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Affiliated Hospital Of Xingtai Medical College, Xingtai, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hospital of Universal Love, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Changzhou NO.2 People's Hospital, Changzhou, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Jiangsu Province Hosipital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Dalian Municipal Central Hospital, Dalian, Liaoning
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang